CLINICAL TRIAL: NCT07393282
Title: A Phase 3, Randomized, Open-Label Study of Linvoseltamab Versus Daratumumab in Participants With Smoldering Multiple Myeloma at High Risk of Developing Multiple Myeloma
Brief Title: A Study to Compare Linvoseltamab and Daratumumab Treatment in High-Risk Smoldering Multiple Myeloma (HR-SMM)
Acronym: LINKER-SMM2
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R5458-HM-24145; 2025-523252-31-00 (EU CTIS Number)
Record Dates: First submitted 2026-01-29; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: High Risk Smoldering Multiple Myeloma (HR-SMM)
Keywords: Linvoseltamab; Multiple Myeloma (MM); B Cell Maturation Antigen (BCMA); Bispecific antibody; Smoldering Multiple Myeloma (SMM); Smoldering Myeloma; HR-SMM; Linozyfic; Darzalex
MeSH Terms: conditions — Multiple Myeloma; Smoldering Multiple Myeloma | interventions — daratumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Linvoseltamab (Experimental)
  Interventions: Drug: Linvoseltamab
- Daratumumab (Active Comparator)
  Interventions: Drug: Daratumumab

INTERVENTIONS:
Drug: Linvoseltamab — Administered per the protocol
  Other Names: REGN5458; Lynozyfic™
  Arms: Linvoseltamab
Drug: Daratumumab — Administered per the protocol
  Other Names: Darzalex Faspro®; Darzalex®
  Arms: Daratumumab

SUMMARY:
This study is researching an experimental drug called linvoseltamab (also called "study drug") compared to another drug called daratumumab, in participants with Smoldering Multiple Myeloma (SMM), who are at a High Risk (HR) of developing active multiple myeloma.

The aim of this study is to find out whether linvoseltamab is better than daratumumab in delaying the development of MM.

The study is looking at several other research questions, including:

* What side effects may happen from taking the study drug
* How much study drug is in the blood at different times
* Whether the body makes antibodies against the study drug (which could make the drug less effective or could lead to side effects)

ELIGIBILITY:
Key Inclusion Criteria:

1. Eastern Cooperative Oncology Group performance status score ≤1
2. SMM diagnosis per IMWG criteria as defined in the protocol
3. Meets HR-SMM criteria by 1 of the risk models as defined in the protocol

Key Exclusion Criteria:

1. Evidence of myeloma-defining events attributable to the underlying plasma cell dyscrasia, as defined in the protocol
2. Diagnosis of systemic light chain amyloidosis, Waldenström macroglobulinemia (lymphoplasmacytic lymphoma), or soft tissue plasmacytoma
3. History of neurodegenerative condition, progressive multifocal leukoencephalopathy or Central Nervous System (CNS) movement disorder
4. History of a seizure within the 12 months of randomization
5. Prior exposure to any approved or investigational treatments directed against a clonal plasma cell disorder (including but not limited to conventional chemotherapies, radiotherapy, immunomodulatory drugs, proteasome inhibitors, anti-CD38 antibodies). Ongoing treatment with other monoclonal antibodies (eg, infliximab, rituximab) or other treatments likely to interfere with study procedures or results, as described in the protocol.

NOTE: Other protocol defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2026-03-25 (Estimated); Primary Completion 2033-07-22 (Estimated); Study Completion 2033-07-22 (Estimated)

PRIMARY OUTCOMES:
Clinical Progression Free Survival (PFS) per International Myeloma Working Group (IMWG) criteria | Up to 5 years
Biochemical PFS per IMWG criteria | Up to 5 years

SECONDARY OUTCOMES:
Achievement of Minimal Residual Disease (MRD) Complete Response (CR) at 10^-5 per IMWG criteria | Up to 12 months
Second PFS (PFS2) | Up to 9 years
Time to death | Up to 9 years
Achievement of Overall Response Rate (ORR) of Partial Response or better (≥PR) per IMWG criteria | Up to 6 months
Best Overall Response (BOR) per IMWG criteria | Up to 5 years
Time to Partial Response or better (≥PR) per IMWG criteria | Up to 6 months
Time to Very Good Partial Response or better (≥VGPR) per IMWG criteria | Up to 5 years
Time to ≥CR per IMWG criteria | Up to 5 years
Achievement of MRD-negativity | Up to 5 years
Sustained MRD-negativity | Up to 5 years
Duration of MRD-negative CR | Up to 5 years
Duration Of Response (DOR) per IMWG criteria | Up to 5 years
Time To Progression (TTP) per IMWG criteria | Up to 5 years
Time to date of initiation of first-line MM therapy | Up to 5 years
Occurrence of Treatment-Emergent Adverse Events (TEAEs) | Up to 5 years
Severity of TEAEs | Up to 5 years
Occurrence of Serious Adverse Events (SAEs) | Up to 5 years
Change from baseline in European Organization for Research and Treatment of Cancer Quality of Life Core Questionnaire 30 (EORTC QLQ-C30) Global Health Status (GHS)/Quality of Life (QoL) scales | Up to 5 years
  The EORTC QLQ-C30 is a 30-item validated questionnaire developed to measure patient-reported QoL using 1 GHS/QoL scale, 5 functioning scales (physical, role, emotional, cognitive and social) and 9 symptom scales / items (fatigue, nausea/vomiting, pain, dyspnea, insomnia, appetite loss, constipation, diarrhea and financial difficulties) among patients with cancer.
  For the functioning scales and global health status / QoL, scores range from 1 = "very poor" to 5 = "excellent" with higher scores indicating better functioning and positive changes from baseline indicate improvement.
Change from baseline in EORTC QLQ-C30 physical scales | Up to 5 years
Change from baseline in EORTC QLQ-C30 role scales | Up to 5 years
Change from baseline in EORTC QLQ-C30 emotional functioning scales | Up to 5 years
Change from baseline in EORTC QLQ-C30 pain scales | Up to 5 years
  The EORTC QLQ-C30 is a 30-item validated questionnaire developed to measure patient-reported QoL using 1 GHS/QoL scale, 5 functioning scales (physical, role, emotional, cognitive and social) and 9 symptom scales / items (fatigue, nausea/vomiting, pain, dyspnea, insomnia, appetite loss, constipation, diarrhea and financial difficulties) among patients with cancer.
  For the 9 symptom scales, scores range from 1 = "not at all" to 9 = "very much" higher scores indicate higher symptom burden and negative changes from baseline indicate improvement.
Change from baseline in EORTC QLQ-C30 fatigue scales | Up to 5 years
Change from baseline in EORTC QLQ- Multiple Myeloma Module 20 (MY20) future perspectives scale | Up to 5 years
  The EORTC QLQ-MY20 is a self -administered instrument to assess QoL in persons with MM. This 20-item questionnaire measures the following domains: symptom scales, including disease symptoms (6 items) and symptoms related to side effects of treatment (10 items); function scale and future perspective (3 items); and body image (1 item)
  A high score for a symptom scale/item represents a high level of symptomatic problem.
Change from baseline in EuroQoL-5 Dimensions, 5-Level Questionnaire (EQ-5D-5L) Visual Analogue Scale (VAS) | Up to 5 years
  The EQ-5D-5L consists of the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The EQ-5D-5L descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: "no problems", "slight problems", "moderate problems", "severe problems" and "extreme problems". The EQ VAS records the participant's self-rated health on a vertical visual analogue scale where the endpoints are labeled "Best imaginable health state" and "Worst imaginable health state".
Functional Assessment of Cancer Therapy (FACIT)- Item Global Population 5 (GP5) responses | Up to 5 years
  FACIT-Item GP5 will be used to assess the patient-reported impact of treatment toxicity that uses a single item "I am bothered by side effects of treatment" on a 5-point scale (0 = not at all, 1 = a little bit, 2 = somewhat, 3 = quite a bit, 4 = very much).
Change from baseline in FACIT- Item GP5 score | Up to 5 years
Concentrations of linvoseltamab in serum over time | Up to 5 years
Occurrence of Anti-Drug Antibody (ADA) to linvoseltamab in serum over the study duration | Up to 5 years
Magnitude of ADA to linvoseltamab in serum over the study duration | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/